CLINICAL TRIAL: NCT02913807
Title: The Utility and Effectiveness of Computer-Assisted, Customized Reconstruction of the Mandible
Brief Title: Traditional Versus Computerized Mandibular Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was ended due to lack of available participants who met criteria.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-34814
Record Dates: First submitted 2016-09-16; First posted 2016-09-26 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Free Tissue Transfer; Mandible Reconstruction; Computerized Customization
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Reconstruction (Placebo Comparator): This cohort will be reconstructed using hand contoured osteotomies and reconstruction bars
  Interventions: Procedure: Hand Contoured Osteotomies and Reconstruction Bars
- Computerized Custom (Experimental): This cohort will be reconstructed using customized computer-modeled titanium locking customized jigs and plates for the osteotomies.
  Interventions: Procedure: Customized Jigs and Plates

INTERVENTIONS:
Procedure: Customized Jigs and Plates — The titanium locking reconstruction plates will be prefabricated based on the preoperative CT scans. Prior to procedure, customized planning for osteotomies will generate the prefabricated jigs.
  Arms: Computerized Custom
Procedure: Hand Contoured Osteotomies and Reconstruction Bars — This will be the traditional method of hand-conjuring the bar and bony sites.
  Arms: Traditional Reconstruction

SUMMARY:
This study will test the accuracy of computerized custom mandibular reconstruction to traditional methods of mandibular reconstruction using a vascularized osteocutaneous fibula flap.

DETAILED DESCRIPTION:
Since the introduction of microvascular repair and the refinement in technique, free tissue transfer has become the gold standard of head and neck reconstruction. Outcomes of free tissue transfer have been also shown to be financially favorable for the healthcare system while improving the quality of life of the patient. The fibula osteocutaneous free flap has established itself as the workhorse for mandibular reconstruction, providing a large amount of bone with an inherently thick cortical stock that makes it an ideal option for creating a new mandible.

Reconstruction of the mandible utilizes a locking reconstruction plate to secure the vascularized bone into position. Paramount to a successful mandibular reconstruction is the accurate contouring of the plate to restore the aesthetic projections and occlusive status of the patient. Computer-assisted, customized reconstruction plate and along with osteotomy jigs (Stryker, CMF) has in-use for mandibular reconstruction. The customized reconstruction plate is similar to the traditional plates except that instead of having to bend them to the proper position, they are manufactured in the properly bent configuration. The stated benefits of such a device would be more accurate contouring resulting in more accurate restorations of the aesthetic projections of the face, better postoperative occlusive status, and a decrease in operative time.

This pilot study is being proposed to determine the variation in mandibular reconstructive outcomes when comparing conventional techniques of manually bent stock reconstruction plates to new methods utilizing pre-surgical planning and customized/patient specific plating. While the customized reconstruction plates and jigs have been studied, there is no head-to-head comparison versus a traditional, hand-bent plate and manually-cut osteotomies. The most commonly used technique at Boston Medical Center is to bend the plates manually, however both techniques are used and can be considered standard of care.

All patients who qualify for reconstruction after tumor ablation, per the investigator institution's tumor board recommendations will be eligible. Recruitment of subjects and enrollment will adhere to IRB requirements. Patients enrolled in the pilot study will be randomized into free hand and computerized groups (N=10 in each arm). All patients will undergo preoperative photographs in standard formats. Those in the free-hand group will undergo mandibular reconstruction using a fibula free flap. The bar will be hand contoured at the time of surgery and the osteotomies will be estimated and performed by hand by the PI per his usual technique. Those undergoing computerized reconstruction will undergo presurgical computerized planning of osteotomies and the reconstruction bar. The remainder of the procedure will go on per the PI's usual procedure for mandibular reconstruction using a fibula free flap. Postoperative treatment between the two groups will not differ from the current standard of care and will occur according to the PI's postoperative protocol. At six months out, patients will undergo CT scanning to evaluate the osteotomy distance and amount of bony contact that is present. Measurements at the outer and inner gaps will be captured as well as the averages between the two. All subjects in each arm will be matched for number of osteotomies and amount of bony defect per procedure. Information regarding length of the total procedure as well as the time specific to the reconstruction and ischemia time (the time from clamping the blood vessels when taking the flap from the leg and then reconnecting them in the neck, and thus re-vascularizing the flap) of the flaps will be collected. Also cephalometric analysis will be performed to evaluate the aesthetic results. See data section for details.

All data collected will be organized and have statistical analysis performed between the two groups. Significant differences will be reported.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will undergo mandibular reconstruction at the Boston Medical Center using a fibula free flap.

Exclusion Criteria:

* Patients under the age of 18
* Prisoners
* Individuals with large lesions that will affect preoperative landmark assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative Osteotomy Gaps as measured via CT measurements (distance=cm) | 6 months postop
  The osteotomy gaps will be measured and an average on each site will be calculated.
Reconstruction Bar | 6 months postop
  The projection and known facial landmarks will be compared suing pre- and post-operative photographs.

SECONDARY OUTCOMES:
Cost and Time | Intraoperative
  The cost-time differences in the OR will be calculated between cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ezzat, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No